CLINICAL TRIAL: NCT01704339
Title: The Role of Qutenza (Topical Capsaicin 8%) in Treating Neuropathic Pain From Critical Ischaemia in Patients With End-stage Renal Failure
Brief Title: Qutenza for Critical Ischaemia in End Stage Renal Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Emma Aitken (Other)
Responsible Party: Sponsor-Investigator, Emma Aitken, Clinical Research Fellow, Renal Surgery, NHS Greater Glasgow and Clyde
Organization: NHS Greater Glasgow and Clyde (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN12RE072; 2012-001586-32 (EudraCT Number)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: End Stage Renal Failure; Neuropathic Pain
Keywords: End stage renal failure; Neuropathic pain; Critical digital ischaemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Neuralgia | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QUTENZA (Experimental): Single treatment with QUTENZA (topical capsaicin 8%) transdermal patch
  Interventions: Drug: QUTENZA

INTERVENTIONS:
Drug: QUTENZA — Single treatment with topical capsaicin 8%
  Other Names: Topical capsaicin 8%

SUMMARY:
Critical ischaemia is pain at rest as the result of poor blood flow and lack of oxygen being delivered to the tissues. It normally affects the hands and feet and can be very debilitating. It is particularly common and difficult to treat in patients with end stage renal failure

Patients with renal failure are often high risk of any operative intervention which might help the pain. Often the only treatment options are painkillers. Unfortunately however, the commonly used painkillers, for example morphine, are known to cause worse side effects in patients with renal failure (drowsiness, confusion etc.

Qutenza (topical capsaicin 8%) is a new treatment made from chilli peppers which is applied to the skin as a patch and works directly at the nerve endings in the skin to prevent pain. It therefore should not have the systemic side effects of other drugs. It has been demonstrated to be beneficial in other painful conditions for example post-shingles pain and nerve pain from HIV. It has never been used for critical ischaemia before.

We propose to investigate the efficacy of Qutenza in treating patients with end stage renal failure and painful ischaemia. We will recruit 20 patients with painful ischaemia and treat them with Qutenza. We will follow them up for 12 weeks and monitor the change in their pain scores.

DETAILED DESCRIPTION:
Peripheral vascular disease is common in end-stage renal failure (ESRF) affecting 24-77% of patients (Stack, 2005). Critical ischaemia (pain at rest caused by insufficient blood supply to a limb) is notoriously difficult to treat in this patient group. Advanced disease and extensive co-morbidities limit surgical revascularisation options of proximal vessels (Blankensteijn et al., 1996) and calciphylaxis (a process of calcification within the small vessels unique to patients with end-stage renal failure) has few effective treatments (Ng & Peng, 2011). Often the only treatment option is symptomatic relief with strong analgesics.

Effective pain relief in patients with end-stage renal failure can be difficult to achieve. The active metabolites of many opiates are renally-excreted and side effects are more common in patients with end-stage renal failure. In particular, confusion and drowsiness limit their use. Similarly drugs commonly used for neuropathic pain, such as gabapentin, have not be investigated in clinical trials in patients with end-stage renal failure (Kurella et al., 1993).

A drug which is not renally excreted, has minimal systemic absorption and does not require dose adjustment in renal failure, is an attractive treatment option for patients with renal failure.

Qutenza (topical capsaicin 8%) is an advanced dermal application system designed for rapid delivery of capsaicin into the skin. The high concentration of capsaicin results in reversible desensitisation of TRPV-1 expressing cutaneous sensory nerve endings and reduction in nerve fibre density in the epidermis (Noto et al., 2009). The resulting pain relief is long-lasting (12 weeks after a single application) (Backonja et al., 2008); Simpson et al., 2008). Previous phase III studies have demonstrated a significant reduction in neuropathic pain in patients with post-herpetic neuralgia (Blonsky et al., 2009) and HIV neuropathy (Noto et al., 2099; Simpson et al., 2008) with a good tolerability profile and it is now licensed for use in treatment of neuropathic pain in these patient groups.

The efficacy and tolerability of Qutenza (topical capsaicin 8%) has been evaluated in over 1,600 patients within clinical trials, with a reduction in pain scores at 8 weeks from 30-32% to 20-24% compared to an active control (capsaicin 0.04%) (Simpson et al., 2008). Patients frequently developed mild irritant symptoms of erythema and itch at the site of application, but significant side effects of blistering were rare occurring in <5%.

Currently Qutenza (topical capsaicin 8%) is not licensed for the treatment of diabetics however there is evidence from a moderate number of diabetics enrolled into clinical trials that Qutenza is both safe and effective in this patient group also. Webster et al, (2011) treated a total of 91 patients with painful diabetic nephropathy and found a 31.5% reduction in mean pain scores during weeks 2-12 post treatment. There was no difference in the incidence of local side effects experienced by diabetics and non-diabetics (Backonja et al, 2011). One patient did develop an ulcer in the area of treatment however it is unclear whether this related to the treatment or not (Webster et al, 2011).

Diabetic patients will be enrolled into this trial due to the frequency of diabetic patients with renal failure and the contributing role of diabetes in small vessel disease leading to critical ischaemia. The distinction between painful diabetic neuropathy and digital critical ischaemia can be difficult to make clinically and it may be that a small proportion of patients recruited for this study also have an element of diabetic neuropathy in addition to their critical ischaemia. In view of the concern with ulceration of the feet in diabetics treated with Qutenza, patients with diabetic neuropathy causing a loss of sensation will be excluded from having their feet treated.

Pain from critical ischaemia is multi-modal and notoriously difficult to treat particularly in patients with established renal failure in whom other analgesic agents are poorly tolerated. A drug such as Qutenza (topical capsaicin 8%) which is not renally excreted, has minimal systemic absorption and does not require dose adjustment in renal failure, is an attractive treatment option for patients with renal failure.

This is a single centre, prospective observational trial evaluating efficacy and tolerability of Qutenza (topical capsaicin 8%) for the treatment of digital critical ischaemia in patients with end stage renal failure.

Primary Objective:

• To evaluate the safety and efficacy of Qutenza (topical capsaicin 8%) in relieving chronic neuropathic pain from digital critical ischaemia in patients with end stage renal failure

Secondary objective:

• To evaluate Quality of Life (QoL) measures in patients with end stage renal failure who have chronic neuropathic pain from critical ischaemia treated with Qutenza (topical capsaicin 8%)

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years old with end stage renal disease on dialysis and critical ischaemia defined as rest pain most days for >3 months

Exclusion Criteria:

* Pre-dialysis
* Hypersensitivity to Qutenza, Emla or any of the excipients
* Broken skin or active ulceration at the site of application
* Severe uncontrolled hypertension (systolic BP >200)
* Proven cardiac event during the preceding 3 months
* Women who are pregnant or breast feeding
* Diabetic neuropathy resulting in a loss of sensation
* Lack of capacity or inability to provide informed consent
* Declines participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Chronic neuropathic pain | 12 weeks
  Chronic neuropathic pain as assessed by Visual Analogue Pain Score

SECONDARY OUTCOMES:
Neuropathic pain | 12 weeks
  As assessed by Brief Pain Inventory
Quality of Life | 6 weeks, 12 weeks
  Assessed using EQ-5D score
Neuropathic pain | 1 week, 6 weeks
  As assesses by Visual Analogue Pain Score
Quality of Life | 12 weeks
  As assessed by Patient Global Impression of Change score
Safety and tolerability | 1 day, 12 weeks
  Skin will be assessed for breaks/ blisters and tolerability including the need for rescue analgesia will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Emma L Aitken, MBChB, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Department of Renal Surgery, Western Infirmary, Glasgow, United Kingdom